CLINICAL TRIAL: NCT01074281
Title: Examination of Patients With Isolated Systolic Hypertonia (ISH) Under Therapy With ENEAS®.
Brief Title: An Observational Study to Examine the Patients With Isolated Systolic Hypertonia (ISH) Under Therapy With Eneas® (NIS ENEAS ISH)
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 084000-501
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
Keywords: Hypertension; Isolated systolic hypertonia; Eneas
MeSH Terms: conditions — Hypertension | interventions — Enalapril; Nitrendipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Enalapril maleate (10 mg) + nitrendipine (20 mg) — The drug was administered as per the Summary of Product Characteristics (SPC)
  Other Names: Eneas

SUMMARY:
This non interventional, multicentric, uncontrolled, prospective, observational study was planned to observe the course of disease in subjects with ISH, who were treated with Eneas.

DETAILED DESCRIPTION:
Isolated systolic hypertonia is an autonomous form of the hypertonia, which in 73% of cases develops from a normal blood pressure (BP) situation. A strict BP control is especially important in older people, since the incidence of the ISH also increases with increasing age. This can be attributed to the elasticity of the vessels reducing with the age. Systolic Hypertension in Elderly Program (SHEP) study has shown ISH to be an independent cardiovascular risk factor.

Eneas is a combination of angiotensin converting enzyme (ACE) inhibitor enalapril maleate (10 mg) and the calcium antagonist nitrendipine (20 mg). Irrespective of the fact as shown in different studies, that calcium-antagonists as also ACE inhibitors have an especially distinctive potential for the degeneration of a left-ventricular hypertrophy (LVH). Examinations like the SYST-EUR-study has demonstrated the high therapeutic potential of the combination of nitrendipine and enalapril in older hypertonia subjects. It was proven in this multicentric, double-blind, randomised and placebo controlled study, that when the additional dose of enalapril (and if necessary diuretics was administered) in subjects with ISH above 60 years under treatment with nitrendipine and in case of not sufficient lowering of BP, the total incidence of cardiac events (heart failure, ischaemic heart disease and sudden heart fall) was reduced by 26% within two years of treatment. As part of the SYST-EUR study, a reduction of the incidence of vascular dementia by 50% was documented in the so-called "Vascular Dementia Project" with standardised psychometric measuring system. This effect was probably attributed not alone to the lowering of BP, but also to the additive ZNS-protective effects of nitrendipine and enalapril.

OBJECTIVES

Primary objective:

* To observe the course of disease in subjects with ISH, who were treated with Eneas. In this case, particular attention was given to achievement of target value in the lowering of the systolic BP value (< 140 mmHg) within a 6 month treatment time period.

Secondary objectives:

* To examine the systolic as well as diastolic BP situation and the total medication, especially medication for the therapy of the ISH across the treatment duration
* To collect the drug security data in the examined subject group under practical conditions

The examination plan of this study included approximately the examinations given below, whereby the time of the individual examinations were subjected exclusively to the clinical requirements and the usual conventions in the centre:

* Examination at the beginning of the treatment (Visit 1)
* Control examination after approximately 3 months (Visit 2)
* Control examination after approximately 6 months (Visit 3)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ISH ≥ 140 / < 90 mmHg
* Subjects who declares his willingness for the participation in the examination
* Subjects aged ≥ 50 years

Exclusion Criteria:

* Subjects who are contraindicated for Eneas

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with ISH ≥ 140 / < 90 mmHg were enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 2065 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Achievement of target BP value of ≤ 140 mmHg | 6 months

SECONDARY OUTCOMES:
Recording of systolic and diastolic BP | 6 months
Recording of the concurrent treatments | 6 months
Side-effects | 6 months

REFERENCES:
- [Result] Trenkwalder, P. (2010). Fixkombination von Enalapril und Nitrendipin bei isoliert systolischer Hypertonie - Wirksamkeit und Verträglichkeit in der täglichen Praxis. Ergebnisse einer multizentrischen, 6-monatigen nichtinterventionellen Studie Perfusion, 23(2), 66.